CLINICAL TRIAL: NCT07221630
Title: Effects of Conventional and Dilutional Ultrafiltration Techniques During Cardiopulmonary Bypass in Pediatric Cardiac Patients
Brief Title: Conventional Ultrafiltration Versus Dilutional Ultrafiltration in Pediatric CPB Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Principal Investigator, Lindsey Stuhm, Certified Clinical Perfusionist, Akron Children's Hospital
Other Study IDs: AkronCH
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: Dilutional Ultrafiltration; Conventional Ultrafiltration; Cardiopulmonary Bypass; C-reactive protein
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample retained for plasma testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional ultrafiltration Group: Conventional ultrafiltration will only have excess effluent removed during cardiopulmonary bypass.
- Dilutional ultrafiltration Group: Dilutional ultrafiltration will have continuous removal of effluent and replacement of this fluid with Plasmalyte.

SUMMARY:
The investigators will be comparing two different filtration methods on cardiopulmonary bypass for pediatric heart surgery patients. Three blood tests will be taken from the patient to compare which filtration method is better at decreasing post-cardiopulmonary bypass inflammation caused by the heart-lung machine.

DETAILED DESCRIPTION:
The study holds promise to evaluate the efficacy of dilutional ultrafiltration (DUF) compared to the currently utilized conventional ultrafiltration method in a prospective randomized controlled trial. A disposable hemoconcentrator is included in the cardiopulmonary bypass circuit which allows for removal of plasma water and solutes with a molecular weight below 65,000 Daltons. Alternatively, dilutional ultrafiltration (DUF) is a process during cardiopulmonary bypass that uses a hemoconcentrator to remove effluent containing inflammatory mediators but also return equal amounts of Plasmalyte to the patient's blood volume through the cardiopulmonary bypass circuit. Plasmalyte is a balanced crystalloid solution that has a similar concentration of electrolytes, osmolality, and pH to human plasma. The "dilutional effect" in DUF is caused by adding Plasmalyte and reducing inflammatory mediators in a patient's entire blood volume while also replacing necessary electrolytes lost during ultrafiltration. The purpose of this study is to examine plasma C-Reactive Protein levels pre-bypass, 12 hours post-bypass, and 24 hours post-bypass comparing the two filtration methods to discover if there is a measurable decrease in postoperative inflammation using dilutional ultrafiltration (DUF) compared to conventional ultrafiltration (CUF). The primary objective of this trial is to evaluate the efficacy of dilutional ultrafiltration (DUF) compared to conventional ultrafiltration (CUF) on cardiopulmonary bypass patients by measuring the outcome of C-Reactive Protein (CRP). The secondary objective is to track postoperative clinical measurements associated with inflammation such as postoperative fluid balance, alveolar arterial gradient, inotrope score, diuretic need, time to negative fluid balance, postoperative length of intubation, and length of ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Males and females less than 5 years of age
* Cardiac operations utilizing CPB
* Cardiac reoperations utilizing CPB

Exclusion Criteria:

* Patients greater than 5 years of age.
* Any active SYSTEMIC noncardiac disease expected to raise patient baseline CRP levels to above normal levels (>1mg/dL). Since CRP levels correlate with the severity of most skin disease, patients with active dermatitis issues on the day of surgery will be excluded from the study. Patients with autoimmune diseases including RA, SLE, IBD (Crohn's disease, ulcerative colitis), Kawasaki disease and patients experiencing active infections will be excluded from the study.
* Any noncardiac disease not well controlled (ex. Asthma not properly controlled with medication, etc.)
* Recent viral illness (ex. Positive COVID/flu test 30 days prior to surgery)
* All patients receive solumedrol (10mg/kg dose) from anesthesia as part of the prebypass protocol. Any patient currently taking steroids will also be excluded from the study
* Non-cardiopulmonary bypass cases (Off pump CoA, Vascular ring surgery, etc.)
* ECMO patients
* Emergent cases

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients having cardiac surgery with cardiopulmonary bypass who meet inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
C-Reactive Protein outcome measure concentration in mg/dL | Baseline measurement
  Measure of acute inflammation in the body
C-Reactive Protein concentration in mg/dL | 12 hours post-bypass
  Measure of acute inflammation in the body
C-Reactive Protein concentration measured in mg/dL | 24 hours post-bypass
  Measure of acute inflammation in the body

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey N Stuhm, MSHS CCP, Principal Investigator — Akron Children's Hospital
Locations (1):
- Akron Children's Hospital, Akron, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Modified and conventional ultrafiltration during pediatric cardiac surgery: clinical outcomes compared. — https://pubmed.ncbi.nlm.nih.gov/17140945/
- See also: Effects of dilutional and modified ultrafiltration in plasma endothelin-1 and pulmonary vascular resistance after the Fontan procedure — https://pubmed.ncbi.nlm.nih.gov/11899192/
- See also: Effect of modified ultrafiltration in high-risk patients undergoing operations for congenital heart disease. — https://pubmed.ncbi.nlm.nih.gov/9768937/
- See also: Hemofiltration increases IL-6 clearance in early systemic inflammatory response syndrome but does not alter IL-6 and TNF alpha plasma concentrations. — https://pubmed.ncbi.nlm.nih.gov/9310806/
- See also: Hemofiltration during cardiopulmonary bypass — https://pubmed.ncbi.nlm.nih.gov/9573598/
- See also: Role of C-Reactive Protein at Sites of Inflammation and Infection. — https://pmc.ncbi.nlm.nih.gov/articles/PMC5908901/